CLINICAL TRIAL: NCT00252486
Title: A Comparison of Omega-3 Fatty Acids vs. Placebo in Children and Adolescents With Bipolar Disorder
Brief Title: Omega-3 Fatty Acids in Children and Adolescents With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00-266
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; Omega-3 Fatty acids
MeSH Terms: conditions — Bipolar Disorder | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flax oil, placebo oil (Placebo Comparator)
  Interventions: Drug: Flax oil

INTERVENTIONS:
Drug: Flax oil — Flax oil and olive oil placebo were analyzed for quality and purity; sufficient bioactivity was confirmed for the flax oil independently at the University of Massachusetts mid-way through the study. Each capsule of omega -3 fatty acid concentrate contained 550 mg of α-linolenic acid (α-LNA) from flax seed oil.A stepped but flexible dose-titration schedule was carried out with doses increased by 1-2 grams at each visit as tolerated, to an attempted total dose of 6 capsules twice per day, as requested by the FDA (up to 6.6 grams of daily α-linolenic acid).
  Other Names: Omega-3 Research Institute, Bethesda, MD

SUMMARY:
The purpose of this study is to test the hypothesis that flax oil, as an omega-3 fatty acid, will be superior to placebo in the maintenance treatment of bipolar disorder in children and adolescents.

Our primary objective was to determine if flax oil is efficacious in the pediatric bipolar population for reducing symptoms of mania and depression. A secondary objective was to examine fatty acid levels as predictors of treatment response and symptom severity. This clinical trial evaluated whether supplementation with flax oil, containing the omega-3 fatty acid alpha-linolenic acid (alpha-LNA), safely reduced symptom severity in youth with bipolar disorder.

DETAILED DESCRIPTION:
Pediatric bipolar disorder is a difficult-to-treat recurrent mental illness characterized by a predominant mood state of irritability, and often mixed, rapid-cycling, and psychotic symptoms. Results of randomized controlled trials of lithium, valproic acid, and antipsychotics for early onset bipolar disorder offer hope of improvement for many, yet also demonstrate need for additional treatment options for those children who do not respond adequately to, or cannot tolerate, a first-line mood stabilizer alone or in combination with an atypical antipsychotic. As popular over-the-counter dietary supplements, omega-3 fatty acids represent an appealing option for treatment in the younger bipolar population as they are likely to be better tolerated and cost less compared with conventional mood stabilizing agents. In addition, they have appeal to parents and adolescents due to their perception as a 'natural' substance and relative lack of systemic side effects. To our knowledge, there are no prospective, randomized, controlled trials of flax oil for the treatment of bipolar disorder or selectively evaluating omega-3 fatty acids in the child and adolescent bipolar population.

Children and adolescents aged 6-17 years with symptomatic Bipolar I or II disorder (n=51), manic, hypomanic, mixed, or depressed, were randomized to either flax oil capsules containing 550 mg alpha-linolenic acid per 1 gram or an olive oil placebo adjunctively or as monotherapy. Doses were titrated to 12 capsules per day as tolerated over 16 weeks. Primary outcomes included changes in the Young Mania Rating Scale (YMRS), Child Depression Rating Scale-Revised (CDRS-R), and Clinical Global Impressions- Bipolar (CGI-BP) ratings using Kaplan-Meier survival analyses. Baseline and end-of-study free fatty acids were measured and examined for change and relevance to effect.

ELIGIBILITY:
Inclusion Criteria:

* male and female outpatients aged 6-17
* DSM-IV diagnosis of bipolar I or II disorder
* currently symptomatic with a CGI of 3 or greater, Y-MRS of 4 or greater, or CDRS-R of 22 or greater
* have failed stabilization with lithium and valproate combined therapy with therapeutic levels documented or are intolerant to these medications
* ability and willingness to provide assent and informed written consent from at least one parent/ legal guardian

Exclusion Criteria:

* mental retardation (IQ less than 70)
* comorbid autism, pervasive developmental disorder, history of substance abuse or positive toxicology screen, or acute post-traumatic stress disorder
* presence of a serious chronic medical illness
* inability to swallow capsules
* pregnant or sexually active without reliable contraception

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2001-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale (YMRS) | EOW 2,4,6,8,10,12,16
Children's Depression Rating Scale (CDRS-R) | EOW 2,4,6,8,10,12,16
Clinical Global Impression - Bipolar Version (CGI) | EOW 2,4,6,8,10,12,16

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Gracious, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Scheffer RE, Kowatch RA, Carmody T, Rush AJ. Randomized, placebo-controlled trial of mixed amphetamine salts for symptoms of comorbid ADHD in pediatric bipolar disorder after mood stabilization with divalproex sodium. Am J Psychiatry. 2005 Jan;162(1):58-64. doi: 10.1176/appi.ajp.162.1.58. PMID 15625202
- [Background] McClellan J, Kowatch R, Findling RL; Work Group on Quality Issues. Practice parameter for the assessment and treatment of children and adolescents with bipolar disorder. J Am Acad Child Adolesc Psychiatry. 2007 Jan;46(1):107-125. doi: 10.1097/01.chi.0000242240.69678.c4. PMID 17195735
- [Background] Nandagopal JJ, DelBello MP, Kowatch R. Pharmacologic treatment of pediatric bipolar disorder. Child Adolesc Psychiatr Clin N Am. 2009 Apr;18(2):455-69, x. doi: 10.1016/j.chc.2008.11.004. PMID 19264273